CLINICAL TRIAL: NCT06827405
Title: Comparison of the Effectiveness of Oral Lactase Enzyme and Lactose Free Formula in the Management of Secondary Lactose Intolerance in Persistent and Severe Persistent Diarrhea
Brief Title: Comparison of the Effectiveness of Oral Lactase Enzyme and Lactose Free Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZUHKARACHI
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Secondary Lactose Intolerance
MeSH Terms: interventions — Lactase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactase enzyme group (Experimental): In this group, 5 drops of lactase enzyme (200 units lactase/drop)/ounce of milk, was added 5-30 minutes before feeding.
  Interventions: Dietary Supplement: Lactase enzyme
- Lactose-free formula feed group (Experimental): In this group, lactose-free formula milk/diet was advised.
  Interventions: Dietary Supplement: Lactose-free formula feed

INTERVENTIONS:
Dietary Supplement: Lactase enzyme — Patients were given 5 drops of lactase enzyme (200 units lactase/drop)/ounce of milk, 5-30 minutes before feeding
  Arms: Lactase enzyme group
Dietary Supplement: Lactose-free formula feed — Patients were advised lactose-free formula milk/diet.
  Arms: Lactose-free formula feed group

SUMMARY:
This study aimed to fill the gaps by comparing the effectiveness of oral lactase enzyme and lactose free formula in the management of secondary lactose intolerance in persistent and severe persistent diarrhea.

DETAILED DESCRIPTION:
Although it is well understood that oral lactase enzyme can play a pivotal role in hastening recovery due to secondary lactose intolerance in persistent diarrhea, there is limited local data available in this regard. If exogenous oral lactase enzyme is found to be more effective, it would help children receive uninterrupted milk and milk-based diet during the diarrheal episode, as the former would aid digestion and absorption of lactose, thus providing the necessary nutrients especially (calcium) and vitamins so vital in this period of rapid growth.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Aged 6-24 months
* Presented with persistent or severe persistent diarrhea due to secondary lactose intolerance
* Patients on formula or mixed feeding, or formula/cow/buffalo milk

Exclusion Criteria:

* Severe acute malnutrition
* Hemodynamic instability (shock)
* Those on oral antibiotics or on excessive juices
* With conditions of malabsorptive states (celiac disease, protein losing enteropathy, or irritable bowel syndrome)

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Resolution of diarrhea | 5 days
  It was labeled on the basis of frequency of stools ≤ 4 and consistency of stools ≤ 5 (Bristol Stool Chart, ideal range 3-5)
Reduction in abdominal pain | 5 days
  A score of ≤ 4, assessed on the basis of faces pain score revised chart (FPS-R), was considered as reduction in pain (a higher score indicating more severe pain)
Lessening in bloating | 5 days
  It was assessed on the basis of a decrease in the abdominal girth (≤ 1) at the umbilicus by a non- stretchable measuring tape
Resolution of nausea/vomiting no perianal rash or only | 5 days
  Decrease in the frequency of nausea/vomiting
Resolution of perianal rash | 5 days
  If no perianal rash or only erythema is seen

SECONDARY OUTCOMES:
Treatment successful | 6 days
  The secondary outcome was treatment success assessed on the basis of all 3 conditions fulfilled, i.e., diarrhea (frequency < 4 stools, consistency < 5) lasting less than 5 days, stool pH > 6, and hospital stays < 5 days.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Ghayas, FCPS, Principal Investigator — Hamdard University Hospital, Karachi; Heena Ghayas, FCPS, Study Director — Ziauddin University Karachi
Locations (1):
- Ziauddin University Hospital, Kemari, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.